CLINICAL TRIAL: NCT05254821
Title: Cell-free Tumor DNA Analysis for Minimal Residual Disease Detection in Patients With Hodgkin Lymphoma
Brief Title: Cell-free Tumor DNA as Minimal Residual Disease in Hodgkin Lymphoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Professor, Federico II University
Other Study IDs: FED-HL-DNA001
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hodgkin Lymphoma
Keywords: ctDNA; Next generation sequencing; Hodgkin lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Molecular analysis identifies residual disease by overcoming the sensitivity of imaging methods and therefore has the potential for integrating with therapy provided by FDG-PET alone. It is a well known fact that tumor DNA circulating in plasma (ctDNA) reflects the mutational profile of tumor cells and can be used to non-invasively detect specific mutations of Hodgkin's lymphoma without the need for microdissecting the histological sample.

DETAILED DESCRIPTION:
A clinical need, not yet met for the Hodgkin lymphoma disease, brings about the early and accurate identification of chemo-refractory patients who require stepping up of treatment as also, patients with good prognosis receiving treatment de-escalation.Molecular methods identify residual disease by overcoming the sensitivity of imaging methods and therefore have the potential to integrate the response to therapy provided by FDG-PET alone.

ctDNA modification from the basal time point to the interim can be used as a predictor of response to the ABVD scheme and as a complement to the interim-PET in the possible variation of the therapeutic schedule.

Clinical data and peripheral blood samples (20 ml in EDTA tubes and 20 ml in Cell-Free DNA BCT tubes) will be collected during the clinico/laboratory visits that are planned as per clinical routine at the time of diagnosis, at each cycle of chemotherapy, at the time of interim PET/CT, at the time of end of treatment PET/CT and during follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years or older
* Documented diagnosis of Hodgkin lymphoma (both classic and nodular predominant lymphocytes subtype) according to 2016 WHO classification
* Willing and able to comply with scheduled study procedures
* Evidence of a signed informed consent
* ECOG performance status 0-2 (or 3, if disease related)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male or female adults 18 years or older with a documented diagnosis of hodgkin lymphoma according to WHO 2016 classification
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of interim ctDNA genotyping | 24 months
  Sensitivity of interim ctDNA genotyping in identifying chemorefractory patients or patients with good prognosis (patients who do not progress after 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Italy